CLINICAL TRIAL: NCT00005158
Title: Segregation/Linkage Analysis for Hypertension
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1030; R01HL028522 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To determine the genetic components of hypertension using a series of simulation experiments designed to determine the power and validity of the then recently developed methods of segregation and linkage analysis.

DETAILED DESCRIPTION:
BACKGROUND:

There are two general hypotheses about the nature of the genetic component of hypertension. A single gene hypothesis visualizes hypertension as a specific disease entity determined by an autosomal dominant or incompletely dominant allele with little environmental effect. A polygenic hypothesis views hypertension as determined by a large number of genetic and environmental factors operating independently with roughly equal contributions. The evidence supporting the single gene hypothesis is based primarily on bimodal and trimodal distributions of blood pressure in the population. It has been suggested that the bimodal or trimodal distributions are the result of ascertainment bias. The evidence supporting the polygenic model is based on several studies where the distribution of blood pressure is unimodal and often skewed toward higher values in both the population and in first degree relatives of hypertensive individuals. These skewed distributions can be approximately normalized using log transformations.

In this study, a particular effort was made to detect major genes. A major gene is said to exist in a particular sample if an appreciable amount of the variability of a trait in that sample is due to segregation of alleles at a single locus. The presence of a major gene does not preclude the existence of other genetic or environmental effects. In the last decade three general models have been proposed to detect the presence of a major gene. The transmission probability model is a general model for the genetic analysis of pedigree data which tests for Mendelian segregation ratios and is a generalization of the traditional methods of segregation analysis. This model has little power to differentiate between single gene and polygenic inheritance although it may be able to detect some kinds of non-single gene transmission. This method has been extended to allow analysis of multivariate traits, testing of a wide variety of hypotheses concerning modes of transmission and various ascertainment corrections. Major genes identified with this model include hypercholesterolemia, dopamine-beta-hydroxylase, and catechol-o-methytransferase.

The mixed model includes both a single locus and a multi-locus component and is designed to distinguish between the two. The model assumes that all transmission from one generation to the next that cannot be accounted for by classical polygenic inheritance is due to segregation of alleles at a single locus. It is ideal for detecting a major gene in the presence of polygenic inheritance provided that no other type of transmission is occurring. This model has been extended to include an environmental correlation among sibs. Major loci identified with this model include PTC, IgE and congenital glaucoma. The unified model is a mixed model with the single locus component parameterized in terms of transmission probabilities, and is a combination of the two previous models. Several research groups have developed methodologies to overcome the computational difficulties presented by this combined model.

DESIGN NARRATIVE:

The study was divided into two parts, the analysis of the methodologies and the application of the methodologies in the genetic analysis of hypertension. In the first part of the study, the power, robustness, and validity of three genetic models of segregation and linkage analysis were considered: the transmission probability model; the mixed model; and the unified model which was also a mixed model with the single locus component parameterized in terms of transmission probabilities. The methods of segregation and linkage analysis found to be most satisfactory were then applied to the analysis of data on five large pedigrees in collaboration with Wright State University and to the analysis of ten large pedigrees ascertained as part of the Bogalusa Heart Study. A determination was made of the effects of partitioning large families into nuclear families and performing segregation and linkage on these nuclear families.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1982-07; Study Completion 1991-06 (Actual)

REFERENCES:
- [Background] Siervogel RM, Weinshilboum R, Wilson AF, Elston RC. Major gene model for the inheritance of catechol-O-methyltransferase activity in five large families. Am J Med Genet. 1984 Oct;19(2):315-23. doi: 10.1002/ajmg.1320190214. PMID 6594929
- [Background] Wilson AF, Elston RC, Siervogel RM, Weinshilboum R, Ward LJ. Linkage relationships between a major gene for catechol-o-methyltransferase activity and 25 polymorphic marker systems. Am J Med Genet. 1984 Nov;19(3):525-32. doi: 10.1002/ajmg.1320190314. PMID 6507499
- [Background] Townley RG, Bewtra A, Wilson AF, Hopp RJ, Elston RC, Nair N, Watt GD. Segregation analysis of bronchial response to methacholine inhalation challenge in families with and without asthma. J Allergy Clin Immunol. 1986 Jan;77(1 Pt 1):101-7. doi: 10.1016/0091-6749(86)90330-1. PMID 3944368
- [Background] Amos CI, Wilson AF, Rosenbaum PA, Srinivasan SR, Webber LS, Elston RC, Berenson GS. An approach to the multivariate analysis of high-density-lipoprotein cholesterol in a large kindred: the Bogalusa Heart Study. Genet Epidemiol. 1986;3(4):255-67. doi: 10.1002/gepi.1370030406. PMID 3744022
- [Background] Asamoah A, Wilson AF, Elston RC, Dalferes E Jr, Berenson GS. Segregation and linkage analyses of dopamine-beta-hydroxylase activity in a six-generation pedigree. Am J Med Genet. 1987 Jul;27(3):613-21. doi: 10.1002/ajmg.1320270314. PMID 3631133
- [Background] Amos CI, Elston RC, Srinivasan SR, Wilson AF, Cresanta JL, Ward LJ, Berenson GS. Linkage and segregation analyses of apolipoproteins A1 and B, and lipoprotein cholesterol levels in a large pedigree with excess coronary heart disease: the Bogalusa Heart Study. Genet Epidemiol. 1987;4(2):115-28. doi: 10.1002/gepi.1370040206. PMID 3108069
- [Background] Wilson AF, Bailey-Wilson JE, Cleton FJ, Elston RC, King MC. Linkage analysis of Dutch families at high risk for breast cancer. Genet Epidemiol Suppl. 1986;1:87-92. doi: 10.1002/gepi.1370030714. No abstract available. PMID 3471674
- [Background] Crowe RR, Noyes R Jr, Wilson AF, Elston RC, Ward LJ. A linkage study of panic disorder. Arch Gen Psychiatry. 1987 Nov;44(11):933-7. doi: 10.1001/archpsyc.1987.01800230013003. PMID 3675131
- [Background] Asamoah A, Wyatt RJ, Julian BA, Quiggins PA, Wilson AF, Elston RC. A major gene model for the familial aggregation of plasma IgA concentration. Am J Med Genet. 1987 Aug;27(4):857-66. doi: 10.1002/ajmg.1320270413. PMID 3480689
- [Background] Wilson AF, Elston RC, Siervogel RM, Tran LD. Linkage of a gene regulating dopamine-beta-hydroxylase activity and the ABO blood group locus. Am J Hum Genet. 1988 Jan;42(1):160-6. PMID 3422127
- [Background] Hill EM, Wilson AF, Elston RC, Winokur G. Evidence for possible linkage between genetic markers and affective disorders. Biol Psychiatry. 1988 Dec;24(8):903-17. doi: 10.1016/0006-3223(88)90225-9. PMID 3233232
- [Background] Tanna VL, Wilson AF, Winokur G, Elston RC. Possible linkage between alcoholism and esterase-D. J Stud Alcohol. 1988 Sep;49(5):472-6. doi: 10.15288/jsa.1988.49.472. PMID 3216652
- [Background] Wilson AF, Cohen JC. Hypotheses for testing deviations from random integration: evidence for nonrandom retroviral integration. Genomics. 1988 Aug;3(2):137-42. doi: 10.1016/0888-7543(88)90144-9. PMID 3224979
- [Background] Wilson AF, Tanna VL, Winokur G, Elston RC, Hill EM. Linkage analysis of depression spectrum disease. Biol Psychiatry. 1989 Jun;26(2):163-75. doi: 10.1016/0006-3223(89)90020-6. PMID 2736265
- [Background] Amos CI, Elston RC, Wilson AF, Bailey-Wilson JE. A more powerful robust sib-pair test of linkage for quantitative traits. Genet Epidemiol. 1989;6(3):435-49. doi: 10.1002/gepi.1370060306. PMID 2753353
- [Background] Tanna VL, Wilson AF, Winokur G, Elston RC. Linkage analysis of pure depressive disease. J Psychiatr Res. 1989;23(2):99-107. doi: 10.1016/0022-3956(89)90001-0. PMID 2585349
- [Background] Bailey-Wilson JE, Elston RC, Wilson AF, Amos CI. A comparison of some sib-pair linkage methods and multiple locus extensions. Prog Clin Biol Res. 1989;329:129-34. No abstract available. PMID 2622941
- [Background] Wilson AF, Elston RC, Sellers TA, Bailey-Wilson JE, Gersting JM, Deen DK, Sorant AJ, Tran LD, Amos CI, Siervogel RM. Stepwise oligogenic segregation and linkage analysis illustrated with dopamine-beta-hydroxylase activity. Am J Med Genet. 1990 Mar;35(3):425-32. doi: 10.1002/ajmg.1320350321. PMID 2309793
- [Background] Bailey-Wilson JE, Dobbins TE. Sib-pair linkage analysis applied to pedigrees with melanoma and dysplastic nevi. Cytogenet Cell Genet. 1992;59(2-3):176-8. doi: 10.1159/000133237. No abstract available. PMID 1737492
- [Background] Wilson AF, Elston RC, Tran LD, Siervogel RM. Use of the robust sib-pair method to screen for single-locus, multiple-locus, and pleiotropic effects: application to traits related to hypertension. Am J Hum Genet. 1991 May;48(5):862-72. PMID 2018038